CLINICAL TRIAL: NCT02479100
Title: An Assessment of the Impact of CONTrast ENhanceD Mammography (CESM) on Patient Management and Comparison With MRI (CONTEND Study)
Brief Title: Contrast Enhanced Spectral Mammography (CESM) Study
Acronym: CONTEND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); GE Healthcare (Industry)
Responsible Party: Principal Investigator, Professor Fiona J Gilbert, Professor of Radiology, Department Head, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RADIOL/2015/CONTEND
Record Dates: First submitted 2015-06-16; First posted 2015-06-24 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Contrast Enhanced Spectral Mammography; Breast; Cancer; Diagnosis; Patient management
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Undergo a CESM (Other): Patients will undergo an experimental Contrast Enhanced Spectral Mammogram (CESM) in addition to standard diagnostic procedures
  Interventions: Diagnostic Test: Contrast Enhanced Spectral Mammogram
- Follow Standard care (No Intervention): Patient will follow standard care pathway.

INTERVENTIONS:
Diagnostic Test: Contrast Enhanced Spectral Mammogram — Undergo a Contrast Enhanced Spectral Mammogram in additional to standard of care
  Arms: Undergo a CESM

SUMMARY:
The aim of this study is to determine if the addition of Contrast Enhanced Spectral Mammography (CESM) to standard diagnostic imaging, results in a decision regarding patient management - discharge, follow-up, surgery or treatment - being made sooner than it would if the patient had followed the standard course of investigations and review.

DETAILED DESCRIPTION:
Women with suspicious breast lesions following mammography and ultrasound will be eligible for the study. Those who consent to participate will be randomised either to receive Contrast Enhanced Spectral Mammography (CESM) in addition to standard care or to receive standard care alone.

Women randomised to receive CESM will undergo the procedure either during the same visit or if necessary on another date within a week. Any additional suspicious lesions detected by CESM will be biopsied along with the original lesion either under ultrasound or x-ray guidance. Biopsy of suspicious lesions is standard care and not part of the research protocol. Those randomised to receive standard care will undergo ultrasound or x-ray guided biopsy of any suspicious lesion identified by ultrasound or mammography.

Results of all biopsies will be discussed at the next multidisciplinary (MDT) meeting where a treatment decision (conservation surgery, mastectomy or neoadjuvent therapy) will be made for those with confirmed disease. MRI will be performed on appropriate women in line with standard practice. Additional disease detected by MRI will be biopsied, either under ultrasound or MRI guidance, if this will influence patient management. The results from these cases will be discussed at the next MDT meeting.

For those women in either arm of the study with benign biopsy results standard care will be followed.

A proforma will be used to record patient pathway, biopsy results and MDT patient management decisions for each case.

For women who received both CESM and MRI, a retrospective review of these images will be made in order to compare diagnostic accuracy. Images from each imaging modality will be read by a different reader for each case. CESM images will be read without the knowledge of MRI results and vice versa. A proforma will be completed by readers to record findings.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to give written informed consent for participation in the study.
* Have a lesion of suspicion 3, 4 or 5 following mammography and ultrasound.

Exclusion Criteria:

* Known or suspected pregnancyBreast implant
* Previous breast cancer
* Known renal impairment
* History of anaphylactoid or anaphylactic reaction to any contrast media
* Contrast media within 24 hours prior to CESM
* Commencement of neo-adjuvant chemotherapy, hormone treatment, radiotherapy or surgery for this episode

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of impact the addition of CESM has on patient management - does this lead to an earlier diagnosis / treatment plan | Retospective analysis at end of data collection period ( approximately I year)
  The pathway of each participant through the diagnostic process will be reviewed at the end of the data collection period to assess whether the addition of CESM resulted in a definitive decision regarding treatment being made earlier than in the usual diagnostic route.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona J Gilbert, FRCR, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

DOCUMENTS (2):
  • Study Protocol (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT02479100/Prot_000.pdf
  • Informed Consent Form (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT02479100/ICF_001.pdf